CLINICAL TRIAL: NCT04837300
Title: Effect of Resisted Sprint and Plyometric Training on Lower Limb Functional Performance in Young Adult Male Football Players. A Randomized Control Trial
Brief Title: Resisted Sprint and Plyometric Training on Lower Limb Functional Performance in Young Adult Male Football Players.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Majmaah University (Other)
Responsible Party: Principal Investigator, Shahnaz Hasan, PhD, Associate Professor, Majmaah University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Majmaah University
Record Dates: First submitted 2021-04-03; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Football Players
Keywords: Strength; Plyometric training; Function performance; Resisted sprint training
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Masking Description: Participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental-1 (Experimental): Resisted Sprint Training
  Interventions: Other: Resisted Sprint Traininig
- Experimental-2 (Experimental): Plyometric Training
  Interventions: Other: Resisted Sprint Traininig
- Control (No Intervention): No Training

INTERVENTIONS:
Other: Resisted Sprint Traininig — The Participants in this group had received plyometrics exercises; double leg jumping, drop jumping, hopping, bounding and hurdling.
  Other Names: Plyometric Training
  Arms: Experimental-1; Experimental-2

SUMMARY:
This study aims to evaluate the short-term effects of resisted sprint training on sprint performance together with lower limb physiological and functional performance in young professional football players.

DETAILED DESCRIPTION:
Ninety collegiate football players were recruited, with a mean age of 20.48 at the university campus. All of which were randomly divided into two experimental groups RST(n=30), PLT (n=30) participated in training for six weeks on alternate days (i.e., three sessions per week) and one control group (n=30) did not train. The control group was instructed to maintain regular activities and avoid any strenuous physical activity during the study. No significant between-group baseline or pre-to-post-training differences in anthropometrics were observed.

Under the Declaration of Helsinki, participants were informed about the study's possible risks and benefits, and all participants have signed informed consent before participation in the study. Ethical sub-committee of College of applied medical science, Majmaah, Saudi Arabia approved this study (Ethics Number: MUREC-Dec.15/COM-2020 / 13-2).

ELIGIBILITY:
Inclusion Criteria:

* Young players aged between 18 and 25 years required frequent sprinting

Exclusion Criteria:

* Current injury to lower limb.
* Surgery affecting lower limb function.
* Any cardio-respiratory diseases.
* Impairments of spine or lower extremities.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 90 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Knee Extensors Strength Test. | After 6 weeks of intervention.
  Pretest and post intervention strength measure.
Sprint Test. | After 6 weeks of intervention.
  Pretest and post intervention sprint measure.
Single-Leg Triple Hop Test. | After 6 weeks of intervention.
  Pretest and post intervention single-leg triple hop measure.

CONTACTS AND LOCATIONS:
Overall Officials: Shahnaz Hasan, PhD, Principal Investigator — Majmaah University
Locations (1):
- Football Playground, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Data has been kept secure with the principal investigator Dr. Shahnaz Hasan and the sub-investigator due to the confidentiality issues.

REFERENCES:
- [Derived] Hasan S, Kandasamy G, Alyahya D, Alonazi A, Jamal A, Unnikrishnan R, Muthusamy H, Iqbal A. Effect of Resisted Sprint and Plyometric Training on Lower Limb Functional Performance in Collegiate Male Football Players: A Randomised Control Trial. Int J Environ Res Public Health. 2021 Jun 22;18(13):6702. doi: 10.3390/ijerph18136702. PMID 34206346